CLINICAL TRIAL: NCT03754114
Title: Brain Oxygen Optimization in Severe TBI (BOOST3): A Comparative Effectiveness Study to Test the Efficacy of a Prescribed Treatment Protocol Based on Monitoring the Partial Pressure of Brain Tissue Oxygen.
Brief Title: Brain Oxygen Optimization in Severe TBI, Phase 3
Acronym: BOOST3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Washington (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, William Barsan, Professor of Emergency Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOOST3; U01NS099046 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Brain Injuries, Traumatic
Keywords: intracranial pressure; hypoxia, brain; critical care; emergency treatment; monitoring, physiologic
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded to the treatment assignment of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICP only (Active Comparator): ICP guided management strategy: Care in the ICU of research participants randomized to this arm will be guided by a monitoring and treatment strategy in which doctors try to prevent high intracranial pressure (ICP) caused by a swollen brain. This strategy is one of two alternative strategies that is currently used in standard care of patients with traumatic brain injury.
  Interventions: Other: ICP guided management strategy
- ICP + PbtO2 (Active Comparator): ICP + PbtO2 guided management strategy: Care in the ICU of research participants randomized to this arm will be guided by a monitoring and treatment strategy in which doctors try to prevent high intracranial pressure (ICP), and also try to prevent low PbtO2 (brain tissue oxygen levels). This strategy is one of two alternative strategies that is currently used in standard care of patients with traumatic brain injury.
  Interventions: Other: ICP + PbtO2 guided management strategy

INTERVENTIONS:
Other: ICP + PbtO2 guided management strategy — In this management strategy, the physiological goal is to avoid ICP from exceeding 22 mm Hg and to avoid PbtO2 dropping below 20 mm Hg. ICP and PbtO2 are monitored using devices inserted into the brain through a hole in the skull. These devices are approved by the US Food and Drug Administration (FDA) and Health Canada for patients with severe TBI. The devices are used in standard care at hospitals participating in this research study. Doctors adjust their treatment choices to try to achieve these ICP and PbtO2 goals. Treatments include kinds and doses of medications and the amount of intravenous fluids given, ventilator (breathing machine) settings, need for blood transfusions, and other medical care. This management strategy is used to guide care for 5 days in this research study.
  Arms: ICP + PbtO2
Other: ICP guided management strategy — In this management strategy, the physiological goal is to avoid ICP from exceeding 22 mm Hg. ICP and PbtO2 are monitored using devices inserted into the brain through a hole in the skull, but PbtO2 is not used to guide care. These devices are approved by the US Food and Drug Administration (FDA) and Health Canada, and are routinely used in patients with severe TBI. Doctors adjust their treatment choices to try to achieve this ICP goal. Treatments include kinds and doses of medications and the amount of intravenous fluids given, ventilator (breathing machine) settings, need for blood transfusions, and other medical care. This management strategy is used to guide care for 5 days in this research study.
  Arms: ICP only

SUMMARY:
BOOST3 is a randomized clinical trial to determine the comparative effectiveness of two strategies for monitoring and treating patients with traumatic brain injury (TBI) in the intensive care unit (ICU). The study will determine the safety and efficacy of a strategy guided by treatment goals based on both intracranial pressure (ICP) and brain tissue oxygen (PbtO2) as compared to a strategy guided by treatment goals based on ICP monitoring alone. Both of these alternative strategies are used in standard care. It is unknown if one is more effective than the other. In both strategies the monitoring and goals help doctors adjust treatments including the kinds and doses of medications and the amount of intravenous fluids given, ventilator (breathing machine) settings, need for blood transfusions, and other medical care. The results of this study will help doctors discover if one of these methods is more safe and effective.

DETAILED DESCRIPTION:
BOOST3 is a randomized clinical trial to determine the comparative effectiveness of two strategies for monitoring and treating patients with traumatic brain injury (TBI) in the intensive care unit (ICU).

When a person has a TBI, their injured brain can swell over a period of hours or days. If the brain swells too much, the pressure in the skull increases and becomes dangerous, causing further injury to the brain. To try to prevent this, doctors usually insert a device, an ICP monitor, into the brain through a hole in the skull of people with severe TBI. An ICP monitor measures the pressure inside the skull. Most doctors agree that it is important to measure and prevent high ICP. Patients with injured brains also suffer additional injury to the brain if the amount of oxygen in the brain gets too low. Some doctors also insert a second device, a PbtO2 monitor, in the brain through the same or a second hole in the skull to measure brain tissue oxygen. A PbtO2 monitor measures how much oxygen is in a small area of the brain near the tip of the monitor. Other doctors think this is unnecessary and unhelpful. Both monitoring devices are approved by the US Food and Drug Administration (FDA) and Health Canada for patients with TBI. Both are commonly used. The ICP and PbtO2 goals guided by these monitors are used to help doctors adjust their treatment choices. Treatments include kinds and doses of medications and the amount of intravenous fluids given, ventilator (breathing machine) settings, need for blood transfusions, and other medical care. Each of these treatment decisions is intended to improve outcomes. However, each treatment decision also involves potential risks. Different treatment decisions may result in different risks. This study will also help doctors better understand these risks. This study is funded by the National Institutes of Health because it answers questions important to the care of patients with TBI.

This study is a two-arm, single-blind, randomized, controlled, phase III, multi-center trial of ICU monitoring and treatment strategies for patients with severe TBI. It will compare the efficacy of ICU care guided by PbtO2 and ICP monitoring versus monitoring of ICP alone in the first 5 days after injury. Only subjects who have severe TBI and require invasive monitoring, according to Brain Trauma Foundation (BTF) and American College of Surgeons-Trauma Quality Improvement (ACS TQIP) guidelines, will be enrolled. All participants in this study will have both ICP monitors and PbtO2 monitors. Half of the participants will be randomized to an arm that includes treatment informed by PbtO2 and ICP, and half will be randomized to an arm that treats only ICP.

The PbtO2 values of those in the ICP only arm will be masked, so that the treating physicians will not be guided by PbtO2 information. Participants in the PbtO2 and ICP arm will have PbtO2 monitored and low measurements treated. Treatments to address physiological goals in both arms will follow a clinical standardization plan. Participants will be followed for 6 months and occurrence of serious adverse events or death will be recorded. Participants will have a follow-up interview to assess their level of recovery approximately 6 months post injury.

To reduce the likelihood of imbalance of important prognostic factors between groups, a covariate-adjusted randomization scheme will be used in this study. Adjustment variables are clinical site and probability of a poor outcome as defined by the IMPACT core model.

ELIGIBILITY:
Inclusion Criteria:

* Non-penetrating traumatic brain injury
* Glasgow Coma Scale (GCS) 3-8 measured off paralytics
* Glasgow Coma Scale motor score < 6 if endotracheally intubated
* Evidence of intracranial trauma on CT scan
* Able to place intracranial probes and randomize within 6 hours of arrival at enrolling hospital
* Able to place intracranial probes and randomize within 12 hours from injury
* Age greater than or equal to 14 years

Exclusion Criteria:

* Non-survivable injury
* Bilaterally absent pupillary response in the absence of paralytic medication
* Contraindication to the placement of intracranial probes
* Treatment of brain tissue oxygen values prior to randomization
* Planned use of devices which may unblind treating physicians to brain tissue hypoxia
* Systemic sepsis at screening
* Refractory hypotension
* Refractory systemic hypoxia
* PaO2/FiO2 ratio < 150
* Known pre-existing neurologic disease with confounding residual neurological deficits
* Known inability to perform activities of daily living (ADL) without assistance prior to injury
* Known active drug or alcohol dependence that, in the opinion of site investigator, would interfere with physiological response to brain tissue oxygen treatments
* Pregnancy
* Prisoner
* On EFIC Opt-Out list as indicated by a bracelet or medical alert

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1094 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | 6 months
  The Glasgow Outcome Scale-Extended (GOS-E) is a global scale for functional outcome, in which higher scores indicate better outcomes. The GOS-E rates patient status into one of eight categories. A GOS-E score of 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery. The categories of severe disability, moderate disability and good recovery are subdivided into a lower and upper category. All injury related disabilities are assessed.

SECONDARY OUTCOMES:
Survival | At discharge from hospital, an average of 19 days
  Survival at discharge from hospital
Total Brain Hypoxia Exposure | Inclusive of up to 5 days of study intervention
  The cumulative area on the time versus brain tissue oxygenation (PbtO2) curve in which PbtO2 is less than 20 mmHg.
Cognition: Rey Auditory Verbal Learning Test | 6 months
  A measure of verbal learning and memory.
Cognition: Trail Making Test Part A+B | 6 months
  A measure of attention, visual-motor tracking and executive functioning.
Emotional Health: Rivermead Post-Concussion Symptom Questionnaire | 6 months
  A measure of the presence and severity of post-concussion somatic, cognitive, and emotional symptoms.
Emotional Health: Brief Symptom Inventory 18 | 6 months
  A measure of psychological distress and psychiatric disorders.
Emotional Health: Satisfaction with Life Scale | 6 months
  A measure of global cognitive judgments of one's life satisfaction.
Functional Status Exam | 6 months
  Change in the activities of every day life as a function of a sudden event or illness

CONTACTS AND LOCATIONS:
Overall Officials: Lori Shutter, MD, Principal Investigator — University of Pittsburgh, Pittsburgh, PA 15260; Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania, Philadelphia, PA 19104; William Barsan, MD, Principal Investigator — University of Michigan, Ann Arbor, MI 48109; Sharon Yeatts, PhD, Principal Investigator — Medical University of South Carolina, Charleston, SC 29425
Locations (54):
- United States (51):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - San Francisco General Hospital, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - NYP Columbia University Medical Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Parkland Hospital, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - WVU Healthcare Ruby Memorial Hospital, Morgantown, West Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (3):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - St. Michaels Hospital, Toronto, Ontario
  - CIUSSS-NIM Hopital du Sacre - Coeur de Montreal, Montreal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after publication on main outcome results paper

REFERENCES:
- [Background] Okonkwo DO, Shutter LA, Moore C, Temkin NR, Puccio AM, Madden CJ, Andaluz N, Chesnut RM, Bullock MR, Grant GA, McGregor J, Weaver M, Jallo J, LeRoux PD, Moberg D, Barber J, Lazaridis C, Diaz-Arrastia RR. Brain Oxygen Optimization in Severe Traumatic Brain Injury Phase-II: A Phase II Randomized Trial. Crit Care Med. 2017 Nov;45(11):1907-1914. doi: 10.1097/CCM.0000000000002619. PMID 29028696
- [Derived] Bernard F, Barsan W, Diaz-Arrastia R, Merck LH, Yeatts S, Shutter LA. Brain Oxygen Optimization in Severe Traumatic Brain Injury (BOOST-3): a multicentre, randomised, blinded-endpoint, comparative effectiveness study of brain tissue oxygen and intracranial pressure monitoring versus intracranial pressure alone. BMJ Open. 2022 Mar 10;12(3):e060188. doi: 10.1136/bmjopen-2021-060188. PMID 35273066
- [Derived] Fiore M, Bogossian E, Creteur J, Oddo M, Taccone FS. Role of brain tissue oxygenation (PbtO2) in the management of subarachnoid haemorrhage: a scoping review protocol. BMJ Open. 2020 Sep 15;10(9):e035521. doi: 10.1136/bmjopen-2019-035521. PMID 32933956
- See also: BOOST3 Study Website — https://siren.network/clinical-trials/boost-3